CLINICAL TRIAL: NCT06537297
Title: The Efficacy and Safety of Intrathecal Pemetrexed With High-dose Furmonertinib Plus Bevacizumab for EGFR-mutant NSCLC Patients With Leptomeningeal Metastases Resistant to Third-generation EGFR-TKIs: A Phase II Study.
Brief Title: Intrathecal Pemetrexed Combined With High-dose Furmonertinib and Beva for EGFR-m NSCLC With Leptomeningeal Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Head of Medical Oncology, Director of Early Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240801
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrathecal Pemetrexed with double Furmonertinib plus bevacizumab (Experimental)
  Interventions: Drug: Intrathecal Pemetrexed and high-dose Furmonertinib plus bevacizumab

INTERVENTIONS:
Drug: Intrathecal Pemetrexed and high-dose Furmonertinib plus bevacizumab — * Intrathecal pemetrexed(50mg) twice a week for 1 week (day 1 and day 5) as induction treatment, then once monthly;
  * Furmonertinib(160mg QD);
  * bevacizumab(5mg/kg，once monthly) until progressive disease.
  Other Names: intrathecal pemetrexed, high-dose furmonertinib, bevacizumab

SUMMARY:
This study aimed to evaluate the efficacy and safety of intrathecal pemetrexed with high-dose Furmonertinib plus bevacizumab for EGFR-mutant non-small cell lung cancer patients with leptomeningeal metastases after resistance to third-generation EGFR-TKIs.

DETAILED DESCRIPTION:
This prospective interventional study aimed to evaluate the efficacy and safety of intrathecal pemetrexed with high-dose Furmonertinib plus bevacizumab for EGFR-mutant NSCLC patients with leptomeningeal metastases after resistance to third-generation EGFR-TKIs.

Approximately 30 EGFR-mutant Non-small cell lung cancer patients with leptomeningeal metastasis or leptomeningeal progression after resistant to third generation EGFR-TKIs were enrolled and treated with intrathecal pemetrexed with high-dose furmonertinib plus bevacizumab. cerebrospinal fluid and blood samples will be collected before and after pemetrexed resistance to analyze molecular mechanisms. Second-generation gene detection will be performed to identify potential resistance mechanisms to pemetrexed. The study is expected to commence recruitment in mainland China in about August 2024. It is expected that the trial will end in April 2026.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
* 2. Age ≥ 18 years.
* 3. Histopathology confirmed Non-small cell lung cancer.
* 4. confirmed or probable leptomeningeal metastases according to EANO-ESMO guidelines or known leptomeningeal metastases progression after third generation of EGFR-TKIs failure.
* 5.Leptomeningeal metastasis (LM) is defined by the presence of typical clinical symptoms, positive cerebrospinal fluid (CSF) cytology, detection of cell-free DNA (cfDNA) in CSF by next-generation sequencing (NGS), or imaging findings consistent with typical meningeal metastases.
* 6.ECOG 0 - 2.
* 7. Predicted survival ≥ 12 weeks.
* 8. Adequate bone marrow hematopoiesis and organ function.

Exclusion Criteria:

* 1. Previously received intrathecal pemetrexed therapy for locally advanced or metastatic disease.
* 2. Subjects who have received any of the following treatments must be excluded: Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
* 3. Presence of spinal cord compression.
* 4. History of other malignant tumors within 2 years.
* 5. Adverse events (except alopecia of any degree) of CTCAE > grade 4 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
* 6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
* 7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
* 8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
* 9. Heart-related diseases or abnormalities
* 10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
* 11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb Furmonertinib due to previous bowel resection.
* 12. Live vaccine was given 2 weeks before the first medication.
* 13. Women who are breastfeeding or pregnant.
* 14. Hypersensitivity to the test drug and the ingredients.
* 15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
LM-overall survival | Time from first subject dose to study completion, or up to last follow up
  LM-OS was defined as the duration from the start of intrathecal pemetrexed to patient death

SECONDARY OUTCOMES:
Extracranial progression-free survival | Time from first dose to the progression of extracranial disease or patient death or last follow up
  Extracranial Progression-Free survival was defined as the duration from the start of intrathecal pemetrexed to the progression of extracranial disease or patient death or last follow up
Clinical response rate | Time from first dose to the improvement of neurological symptoms and KPS score
  Clinical Response Rate was defined as the ratio of the patient whose neurological symptoms and KPS improved according to the criteria of clinical response
Adverse events (AEs) | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China